CLINICAL TRIAL: NCT02428959
Title: Prospective Study to Assess the Diagnostic Utility of Amyl Nitrite in Patients With Suspected Achalasia Undergoing High Resolution Esophageal Manometry (HREM)
Brief Title: Diagnostic Utility of Amyl Nitrite in Patients With Suspected Achalasia Undergoing High Resolution Esophageal Manometry (HREM)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00029912
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Dysphagia; Achalasia
Keywords: Amyl Nitrite; High Resolution Manometry
MeSH Terms: conditions — Deglutition Disorders; Esophageal Achalasia | interventions — Amyl Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amyl Nitrite (Experimental): Amyl nitrite is the chemical compound with the formula C5H11ONO. It relaxes vascular smooth muscle.The method of administration is via inhalation with onset of action within of 30 seconds and ends 2-3mins. In a study by Dodds et al., amyl nitrite is used as part of radiologic esophagram test in order to distinguish patients with pseudoachalasia from those with idiopathic achalasia since amyl nitrite has transient effect on the lower esophageal sphincter (LES). The study revealed that the LES pressure in achalasia patient decreases substantially in response to amyl nitrite with the measurable increase in LES diameter of 3 mm to an average of 4.6m. In contrast, amyl nitrite does not relax the LES segment in pseudoachalasia and has no change in LES diameter. Thus, the investigators anticipate amyl nitrite inhalation will be beneficial at the LES during HREM.
  Interventions: Drug: Amyl Nitrite

INTERVENTIONS:
Drug: Amyl Nitrite — Amyl nitrite is the chemical compound with the formula C5H11ONO. It relaxes vascular smooth muscle; decreases venous ratios and arterial blood pressure; reduces left ventricular work; decreases myocardial oxygen consumption. The method of administration is via inhalation with onset of action within of 30 seconds and ends 2-3mins. In a study by Dodds et al., amyl nitrite is used as part of radiologic esophagram test in order to distinguish patients with pseudoachalasia from those with idiopathic achalasia since amyl nitrite has transient effect on the lower esophageal sphincter (LES). The study revealed that the LES pressure in achalasia patient decreases substantially in response to amyl nitrite with the measurable increase in LES diameter of 3 mm to an average of 4.6m. In contrast, amyl nitrite does not relax the LES segment in pseudoachalasia and has no change in LES diameter. Thus, the investigators anticipate amyl nitrite inhalation will be beneficial at the LES during HREM.

SUMMARY:
This research is being done to see if a study drug called amyl nitrite can be helpful with diagnosing different disorders affecting the lower esophageal sphincter in patients with dysphagia (difficulty swallowing foods) undergoing high resolution esophageal manometry (HRM).

Dysphagia may be one of the symptoms of a condition known as idiopathic achalasia. Achalasia is a disorder of the esophagus, the tube that carries food from the mouth to the stomach. This affects the ability of the esophagus to move food toward the stomach. Pseudoachalasia is a secondary form of achalasia, which has very similar symptoms but is caused by different reasons. Because the treatments for achalasia and pseudoachalasia are different, it is important to correctly diagnose each condition. At this time, there is no way to distinguish the two with the current tests used at Johns Hopkins.

Amyl nitrite relaxes vascular smooth muscle and has been studied previously as a potential means to separate achalasia from pseudoachalasia. Amyl nitrite is approved by the Food and Drug Administration (FDA) for the treatment of cardiac angina. It is not approved for use in motility testing and its use in this study is considered investigational. Investigators hope that the results from the proposed study could have significant clinical implications for patient management by helping doctors distinguish between achalasia and pseudoachalasia and allow them to choose appropriate treatment.

Patients with dysphagia (difficulty swallowing foods) undergoing routinely scheduled high resolution esophageal manometry (HRM) may join this study.

DETAILED DESCRIPTION:
A single center, prospective study at a tertiary-care referral center (JHH). All patients will be provided with informed consent to undergo HRM with provocation as part of routine care to evaluate dysphagia symptoms or evaluation of known achalasia. All procedures will be performed as part of routine care and therefore no procedures will be performed for the purposes of research specifically.

Primary Objective: To determine the diagnostic advantage of the addition of the provocative amyl nitrite test in patients with dysphagia undergoing high resolution esophageal manometry (HRM)

Secondary Objective:

1. Measure change of LES pressure after amyl nitrite inhalation in patients with dysphagia undergoing high resolution esophageal manometry (HRM)
2. To assess the ability of amyl nitrite inhalation to differentiate achalasia from pseudoachalasia
3. To assess the ability of amyl nitrite inhalation to differentiate partial fundoplication-related dysphagia versus that due to recrudescence of achalasia in patients who have undergone a prior myotomy.
4. To assess the ability of amyl nitrite inhalation to differentiate post-fundoplication dysphagia from a newly diagnosed motility disorder in patients who have undergone a fundoplication for gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old
* symptoms of dysphagia or a known history of achalasia

Exclusion Criteria:

* Patients with comorbidity and contraindications to use of amyl nitrite inhalation: Glaucoma, Recent head trauma or cerebral hemorrhage, Hypotension, Concurrent use of nitrite, Pregnancy, Aortic stenosis, Patients with increased intracranial pressure, Caution in patients with coronary artery disease, Pulmonary hypertension
* Non-English speakers
* Patients <18 years old
* Those who lack capacity to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Measure LES pressure after amyl nitrite inhalation in patients with dysphagia undergoing high resolution esophageal manometry (HRM) | 3 months

SECONDARY OUTCOMES:
Measure Blood Pressure and Heart Rate at baseline and after administration of amyl nitrite | 1 month
Number of Participants with Adverse Events with amyl nitrite inhalation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Stein, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States